CLINICAL TRIAL: NCT05816174
Title: Child and Parent Emotion-related Risk and Resilience Factors Associated With the Transition From Acute to Chronic Pain After Surgery: A Prospective Longitudinal Study
Brief Title: Longitudinal Study of Chronic Postsurgical Pain in Children and Adolescents
Status: Recruiting | Type: Observational
Sponsor: Helen Koechlin (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Helen Koechlin, Principal Investigator, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Other Study IDs: LORRIS
Record Dates: First submitted 2023-03-30; First posted 2023-04-18 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Chronic Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic postsurgical pain is defined as pain that develops or intensifies following a surgical procedure. After major surgery, around 20% of children and adolescents develop chronic postsurgical pain, and, as part of it, negative consequences on their quality of life. Emotion-related factors such as the variability of emotions, how emotions are regulated, and how well someone is able to differentiate between different emotions have in part been studied in other types of chronic pain. To date, no study examined emotion-related factors in the development and maintenance of chronic postsurgical pain. This observational study includes five assessment time points, one before and four after major surgery, with the goal to identify emotion-related factors that increase or decrease the risk for the development of chronic postsurgical pain.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged between 8 and 18 years
* Planned orthopedic surgery requiring in-patient care in one of the participating children's hospitals
* Able to read and understand German

Exclusion Criteria:

* Serious comorbid health condition (e.g., cancer, severe neurological impairment, chronic illness requiring daily medication)
* Prior major orthopedic surgery (e.g., prior spine surgery)
* Parent/caregiver and child not able to read and understand German

Ages: 8 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants between the ages of 8 and 18 years who have a planned orthopedic surgery in one of the participating hospitals will be approached. Participating hospitals are large Swiss university children's hospital.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Chronic postsurgical pain | 3 months
  Chronic postsurgical pain as defined by the International Association for the Study of Pain, i.e.: greater than minimal pain (pain intensity ≥ 3) on more than 50% of a 7 days period, and impairment in health-related quality of life (score of < 74.9 on the Pediatric Quality of Life Inventory, PedsQL). This results in a binary outcome: chronic postsurgical pain yes vs no.
Pain trajectories | 12 months
  Description of pain trajectories over time, i.e., from baseline through FU3 (at 12 months after surgery). We will estimating group-based trajectory models using participants' Numeric Rating Scale (NRS) values of pain intensity at each time point. Higher ratings on the numeric rating scale indicate more pain.
Emotion-related trajectories | 12 months
  Description of emotion-related trajectories over time, i.e., from baseline through Follow-up 3 (at 12 months after surgery). We will estimating group-based trajectory models using participants' Visual Analogue Scale (VAS) values of emotional state to calculate emotion differentiation, emotion variability, and emotion regulation at each time point and describe changes over time. Higher values for emotional variability indicate broader range of emotional fluctuations around an individual's mean. Emotion differentiation will be calculated by means of intraclass correlations, with high consistency across predefined episodes indicate poorer differentiation.

SECONDARY OUTCOMES:
Physical activity | 3 months
  Number of steps taken by patients per day, as measured by an ambulatory, non-invasive activity-monitoring device worn around the wrist. Higher number of steps taken suggests more physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Koechlin, PhD, Principal Investigator — University Children's Hospital, Zurich
Locations (3):
- Switzerland (3):
  - University Children's Hospital Basel, Basel
  - University Children's Hospital Zurich, Zurich
  - University Hospital Balgrist, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hochreuter J, Dreher T, Hasler CC, Canonica S, Locher C, Held U, Rabbitts J, Koechlin H. Longitudinal Resilience and Risk Factors in Pediatric Postoperative Pain (LORRIS): Protocol for a Prospective Longitudinal Swiss University Children's Hospitals-Based Study. BMJ Open. 2024 Mar 28;14(3):e080174. doi: 10.1136/bmjopen-2023-080174. PMID 38548365